CLINICAL TRIAL: NCT02907554
Title: Effects of Cyclosporine a Pretreatment of Deceased Donor on Kidney Graft Function: a Randomized Controlled Trial
Brief Title: Cyclosporine a Pretreatment and Kidney Graft Function
Acronym: Cis-A-Rein
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: University Hospital, Estaing (Other); Centre Hospitalier Universitaire de Nice (Other); Groupe Hospitalier Pitie-Salpetriere (Other); Centre Hospitalier Universitaire de Nīmes (Other); University Hospital, Montpellier (Other); Hôtel Dieu (Nantes) (Unknown); Poitiers University Hospital (Other); University Hospital, Toulouse (Other); Hôpital de la Timone (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RBHP_2014_CONSTANTIN; 2014-003544-12 (Other: 2014-003544-12)
Record Dates: First submitted 2016-09-05; First posted 2016-09-20 (Estimated); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Brain Death; Kidney Transplantation
Keywords: Preconditioning; Tissue and organ procurement; Cyclosporine A; Kidney transplantation; Delayed graft function
MeSH Terms: conditions — Brain Death; Delayed Graft Function | interventions — Cyclosporine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (Placebo Comparator): control group receives a placebo
  Interventions: Drug: Placebo
- intervention group (Experimental): the intervention group receives 2.5 mg/kg of cyclosporine
  Interventions: Drug: cyclosporine A

INTERVENTIONS:
Drug: cyclosporine A — the intervention group receives 2.5 mg/kg of cyclosporine
  Arms: intervention group
Drug: Placebo — control group receives a placebo
  Arms: control group

SUMMARY:
Organ donors included in the study are randomized to a control group or an intervention group receiving 2.5 mg/kg of cyclosporine A before organ procurement. Harvested kidneys from these patients are transplanted to chronic kidney insufficiency patients. According to the pretreatment of the transplant, delayed graft function during the first week was evaluated as well as kidney function at different timepoints and mortality during the first year after transplantation.

DETAILED DESCRIPTION:
Organ donors included in the study are randomized to a control group receiving a placebo or an intervention group receiving 2.5 mg/kg of cyclosporine A before organ procurement. In the operating theater organs are harvested. Thereafter, harvested kidneys from these patients are transplanted to chronic kidney insufficiency patients. The management of transplanted patients is performed as usual. According to the pretreatment of the transplant, delayed graft function during the first week (need of at least one dialysis session) was evaluated as well as kidney function at different timepoints (slow graft function, estimated creatinine clearance on day 3 and 7, acute and chronic graft rejection), length of hospital stay and mortality during the first year after transplantation.

ELIGIBILITY:
Inclusion Criteria:

For organ donors:

* Male and females aged 18 to 80 years
* Brain death

Inclusion criteria for organ recipients:

* Male and females aged 18 to 80 years
* Indication of kidney transplantation
* Informed consent

Exclusion Criteria:

For organ donors:

* Contra-indication for multiorgan procurement (infections, cancer, etc)
* Preexistent chronic renal failure.
* Refusal for organ procurement by the donor (confirmed by the French national register or reported by the next-of-kin).

Exclusion criteria for organ recipients:

* Need for a double kidney transplantation.
* Need for a multiorgan transplantation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 648 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2022-04-10 (Actual); Study Completion 2023-04-03 (Actual)

PRIMARY OUTCOMES:
Percentage of delayed graft function defined by a need of at least one hemodialysis session | within the 7 days following renal transplantation.

SECONDARY OUTCOMES:
Percentage of slow graft function defined by a urine output < 1000 ml | at on 1 day after transplantation
Percentage of slow graft function defined by a decrease in plasma creatinine concentration of less than 30% or 70% | at day 3 and 7 after transplantation
Postoperative evolution of estimated creatinine clearance | at day 3 and 7
Percentage of acute and chronic graft rejection | during the first year after transplantation
Percentage of primary graft dysfunction | during the first year after transplantation
hospital length of stay | at day 1
  after transplantation
Mortality | during the first year after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Carole ICHAI, Principal Investigator — CHU NICE
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Orban JC, Fontaine E, Cassuto E, Baumstarck K, Leone M, Constantin JM, Ichai C; AzuRea network. Effects of cyclosporine A pretreatment of deceased organ donors on kidney graft function (Cis-A-rein): study protocol for a randomized controlled trial. Trials. 2018 Apr 17;19(1):231. doi: 10.1186/s13063-018-2597-4. PMID 29665840